CLINICAL TRIAL: NCT02843178
Title: Coupons for Healthy Intake Using Variable Economic Strategies (CHIVES)
Brief Title: Designing Food Voucher Programs to Reduce Disparities in Healthy Diets
Acronym: CHIVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 36763
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases
Keywords: nutrition; food security; behavioral economics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1: distributed, targeted vouchers (Experimental): Participants receive four $5 vouchers each valid for a subsequent week of the month (i.e., one voucher valid for week 1 only, a second for week 2 only, a third for week 3 only, and a fourth for week 4 only), starting in month 1 and continuing every month through month 6. The voucher is restricted to pay for fruits and vegetables.
  Interventions: Behavioral: Vouchers
- 2: lump sum, targeted vouchers (Active Comparator): Participants receive four $5 vouchers each valid for an entire month, starting in month 1 and continuing every month through month 6. The voucher is restricted to pay for fruits and vegetables.
  Interventions: Behavioral: Vouchers
- 3: distributed, untargeted vouchers (Active Comparator): Participants receive four $5 vouchers each valid for a subsequent week of the month (i.e., one voucher valid for week 1 only, a second for week 2 only, a third for week 3 only, and a fourth for week 4 only), starting in month 1 and continuing every month through month 6. The voucher can pay for any food but not tobacco, alcohol or prepared foods.
  Interventions: Behavioral: Vouchers
- 4: lump sum, untargeted vouchers (Active Comparator): Participants receive four $5 vouchers each valid for an entire month, starting in month 1 and continuing every month through month 6. The voucher can pay for any food but not tobacco, alcohol or prepared foods.
  Interventions: Behavioral: Vouchers

INTERVENTIONS:
Behavioral: Vouchers — A voucher is given that can be used at the cashier of participating grocery stores, corner stores, and farmer's markets, enabling a participant to have the voucher's value subtracted from their grocery bill.

SUMMARY:
Improving diets through increased food and vegetable (F&V) consumption significantly reduces the risk of cardiovascular disease (CVD). Programs increasing the accessibility and affordability of F&Vs among low-income Americans have been hindered by the food consumption cycle associated with poverty: the tendency to over-consume calories shortly after receiving funds at the beginning of each month, draining the budget for F&V purchases, or for all food purchases, by month's end. An emerging theory about dietary behavior suggests that providing funds for food in smaller installments distributed throughout the month will smooth the consumption cycle and improve healthy eating-counteracting the tendency to respond to lump sum, once-monthly funding installments by purchasing calorie-dense foods immediately after funds are received. The theory also suggests that funds targeted toward specific healthy foods (e.g., F&Vs) will improve diets more than untargeted funds, despite the inconvenience of utilizing targeted funds. We will rigorously test both hypotheses in a real-world setting by comparing alternative approaches for delivering food purchasing vouchers. We have established and tested the infrastructure to provide vouchers accepted by numerous food sellers (e.g., supermarkets, corner shops) in low-income neighborhoods. Leveraging this infrastructure, we will conduct a randomized trial with a two-by-two factorial design, comparing $20 of vouchers valid for one month to four $5 vouchers each valid for a sequential week of the month (lump sum versus distributed funding), and comparing vouchers restricted to F&V purchases to vouchers redeemable for any food (targeted versus untargeted funding). Low-income adults (N=288) recruited through our community partners will be randomized to one of four 6-month interventions: monthly targeted, monthly untargeted, weekly targeted, or weekly untargeted vouchers. Participants will be assessed through efficient verbal 24-hour dietary recalls validated among low-literacy populations, to determine daily consumption of F&Vs and metrics of overall dietary quality at months 0, 6 and 12 (6 months after vouchers end). Additional surveys will identify moderators and mediators of dietary improvement.

DETAILED DESCRIPTION:
Participants for the trial will be recruited via advertisements at community sites including primary care clinics, housing assistance sites, and soup kitchens in the city of San Francisco. Recruitment materials will direct interested individuals to attend one of the study information sessions at a 'store front' site in San Francisco for an initial screening evaluation by the study staff, and a study orientation session to detail the study purpose, procedures, and participant rights. The orientation sessions will consist of a 60-minute session at a centrally-located room. After the orientation session, participants will be invited to sign a consent form, complete the baseline assessment, and be randomized to one of the four intervention conditions in a 1:1:1:1 allocation. We will use permuted block randomization so that sample sizes in each intervention group are nearly equal. Allocation sequence will be concealed prior to assignment; staff for sequence generation, allocation concealment, and implementation will be separate.

Those agreeing to participate will sign a written consent form after the study orientation and before randomized to one of four voucher conditions, as part of our 2-by-2 study design: (1) vouchers targeted to fruits and vegetables and valid for sequential weeks of the month; (2) vouchers targeted to fruits and vegetables and valid over the entire month; (3) vouchers applicable to any food and valid for sequential weeks of the month; and (4) vouchers applicable to any food and valid over the entire month. Half of participants will receive a blue voucher valid for any food (not tobacco, alcohol, or prepared foods), while the other half will receive a green voucher valid only for qualified fruits and vegetables (fresh or frozen fruits, vegetables, or herbs without added sugars or fats, to correspond to the eligibility guidelines of existing voucher programs). All vouchers will have the same individual value ($5), but one half of participants will receive four vouchers that are each valid for the whole month (a lump sum payment of $20), while the other half will receive four vouchers that are each valid for one sequential week of the month, as labeled on the voucher (a distributed payment of $5 per week). Therefore, all intervention groups will be balanced on time and attention from study staff, as well as effort to obtain the vouchers. By having all vouchers in small increments of $5, we minimize the need for a large voucher to be spent all at once, reducing the risk of food spoilage affecting intervention effectiveness. Having all vouchers be worth the same value also simplifies processing of the voucher at the level of the food vendor. We have specifically designed the monetary amounts of the trial to be sufficient for achieving nutritional goals (the Healthy People 2020 goal of consuming 1.4 cups of fruits and vegetables per day), but not be unduly large so as to be coercive to low-income populations.

Vouchers will be mailed to each participant toward the end of the month prior that the vouchers were valid for, i.e. vouchers for March 2017 will be mailed at the end of February 2017. Vouchers will be prepared following the guidelines in the Trial Protocol.

To redeem vouchers, participants present the voucher to a cashier, and sign and date the voucher at the time of redemption. The cashier processes the voucher just as they processes vouchers for the Women, Infants and Children's program or manufacturer's coupons, and the vendor then submits the redeemed voucher for payment (the financial infrastructure is handled by the San Francisco General Hospital Foundation). The names of the vendors who will accept the vouchers are printed on each voucher, along with their address and business hours. All voucher rules will be reviewed with participants during the orientation session. We will continue routine meetings with the neighborhood food vendors' managers to ensure continued active participation and correct usage of the vouchers.

Following informed consent, participants will complete a baseline survey and a 24-hour dietary recall before being randomized to one of the four study conditions. The recall includes three distinct passes to obtain a participant's food intake during the previous 24 hours-a quick list, a detailed description, and a review-including foods obtained at home and away from home, and including bartered, foraged, food pantry and other non-purchased items. Participants are provided standard 2-dimensional booklets for reference to portion sizes. Our research assistants are blinded to the participant's intervention arm and skilled in guiding dietary recalls among diverse participants in a non-judgmental, comprehensive manner. The baseline recall will be conducted in person at the store front site; subsequent recalls will be conducted over telephone. Recalls will be performed during week 1 and week 4 of the month-0 (baseline), month-6, and month-12 assessments. Two recalls each will be done during week 1 (one weekday and one weekend) and two during week 4 (one weekday and one weekend) of the assessment months. This minimizes the number of recalls required to capture intra-person variation in diet between weekdays and weekends, while simultaneously capturing the monthly consumption cycle among participants (the key hypothesized mediator for the lump sum vs. distributed voucher effect).

In addition to dietary recalls, research assistants will orally administer surveys to prevent literacy-based biases, consistent with recent Institute of Medicine recommendations. These 20-minute surveys will be conducted at months 0, 6, and 12 and will cover attitudes and preferences regarding the vouchers and fruits and vegetables generally, shopping patterns, food expenditures, household environment, and food insecurity.

Each participant will receive vouchers for a total of 6 months. The participants will then be tracked by the recruitment/retention coordinator through brief telephone contact monthly to ensure retention until they complete the month 12 survey and dietary recall (6 months after the end of the intervention), after which they are discharged from the study.

In addition to participants who receive the vouchers, we will also conduct a brief survey with managers of the ten stores who have signed memos of understanding with the City of San Francisco and San Francisco General Foundation to accept the vouchers. The managers will be given informed consent forms to consider participating in a post- intervention survey. The paper-based vendor survey will be hand-delivered to vendors' managers to assess: (i) whether managers have any difficulties with the voucher system and whether those difficulties are at the point of sale, at the point of reimbursement, and/or when answering questions to customers about the vouchers; (ii) what if any activities were used by vendors to promote fruit and vegetable purchases during the voucher trial period; (iii) what if any activities they had engaged in to sell more fruits and vegetables; and (iv) a free text entry to elicit what changes vendors would propose to the voucher system in future

ELIGIBILITY:
Inclusion Criteria: age ≥21 years; household income <250% of the federal poverty level; has regular access to a phone; understands English sufficiently to provide informed consent; a resident of the City of San Francisco as defined by official municipal boundaries; willing to be randomized. Exclusion Criteria: participating in a diet including any other dietary or nutrition study; currently has diagnosed cancer or congestive heart failure; is pregnant; planning to move in the next year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2016-12; Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Basu, MD, PhD, Principal Investigator — Stanford University; Hilary K Seligman, MD, MS, Principal Investigator — University of California, San Francisco; Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- CHIVES Study Office, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White JS, Basu S. Does the benefits schedule of cash assistance programs affect the purchase of temptation goods? Evidence from Peru. J Health Econ. 2016 Mar;46:70-89. doi: 10.1016/j.jhealeco.2016.01.005. Epub 2016 Jan 29. PMID 26874596
- [Background] Whittle HJ, Palar K, Hufstedler LL, Seligman HK, Frongillo EA, Weiser SD. Food insecurity, chronic illness, and gentrification in the San Francisco Bay Area: An example of structural violence in United States public policy. Soc Sci Med. 2015 Oct;143:154-61. doi: 10.1016/j.socscimed.2015.08.027. Epub 2015 Aug 20. PMID 26356827
- [Background] Seligman HK, Bolger AF, Guzman D, Lopez A, Bibbins-Domingo K. Exhaustion of food budgets at month's end and hospital admissions for hypoglycemia. Health Aff (Millwood). 2014 Jan;33(1):116-23. doi: 10.1377/hlthaff.2013.0096. PMID 24395943
- [Result] Basu S, Gardner CD, White JS, Rigdon J, Carroll MM, Akers M, Seligman HK. Effects Of Alternative Food Voucher Delivery Strategies On Nutrition Among Low-Income Adults. Health Aff (Millwood). 2019 Apr;38(4):577-584. doi: 10.1377/hlthaff.2018.05405. PMID 30933599

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Started | 86 | 90 | 92 | 91
Completed | 78 | 82 | 85 | 87
Not Completed | 8 | 8 | 7 | 4
Not completed — Lost to Follow-up | 8 | 8 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers | Total
Number analyzed (Participants) | 86 | 90 | 92 | 91 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.1) | 50.7 (13.4) | 52.4 (14.1) | 50.9 (13.5) | 51.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 61 | 57 | 234
  Male | 30 | 30 | 31 | 34 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 13 | 15 | 56
  Not Hispanic or Latino | 72 | 76 | 79 | 76 | 303
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4 | 1 | 9
  Asian | 17 | 17 | 13 | 14 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 24 | 24 | 21 | 21 | 90
  White | 35 | 28 | 40 | 39 | 142
  More than one race | 2 | 8 | 8 | 7 | 25
  Unknown or Not Reported | 6 | 11 | 5 | 8 | 30
Region of Enrollment [Number; unit: participants]
  United States | 86 | 90 | 92 | 91 | 359
SNAP participation [Count of Participants; unit: Participants] — Participants reporting current active participation in the federal Supplemental Nutrition Assistance Program (SNAP).
  Participants | 22 | 26 | 26 | 25 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Cup-equivalents of Fruit and Vegetable Intake From Baseline to Month 6
Description: Fruit and vegetable intake (measured in Cup-equivalents) at the end of month 6 of the trial, assessed by 24-hour dietary recall
Time Frame: Baseline and Month 6
Measure: Mean (95% Confidence Interval); unit: Change in Cup-equivalents, mo 0 to mo 6
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
Change in Cup-equivalents, mo 0 to mo 6 | 0.18 [-0.004 to 0.36] | 0.08 [-0.09 to 0.26] | 0.09 [-0.09 to 0.26] | 0.04 [-0.13 to 0.21]

2. Secondary Outcome: Change in Cup-equivalents of Fruit and Vegetable Intake From Baseline to Month 12
Description: Fruit and vegetable intake (measured in Cup-equivalents) at the end of month 12 of the trial (6 months after voucher program has ended), assessed by 24-hour dietary recall.
Time Frame: Baseline and Month 12
Measure: Mean (95% Confidence Interval); unit: Change in Cup-equivalents, mo 0 to mo 12
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
Change in Cup-equivalents, mo 0 to mo 12 | 0.0316 [-0.1529 to 0.2161] | 0.0180 [-0.1655 to 0.2015] | -0.0849 [-0.2689 to 0.0991] | 0.2112 [0.0315 to 0.3909]

3. Secondary Outcome: Change in Healthy Eating Index From Baseline to Month 6
Description: Healthy Eating Index (a composite metric of nutrition quality) estimated from 24-hour dietary recall. The scores range from 0 to 100. An ideal overall Healthy Eating Index score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans (DGA).
Time Frame: Baseline and Month 6
Measure: Mean (95% Confidence Interval); unit: change in Index from mo 0 to mo 6
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
change in Index from mo 0 to mo 6 | 1.2 [-0.9 to 3.3] | 0.7 [-1.3 to 2.7] | 2.1 [0.1 to 4.0] | -0.3 [-2.3 to 1.7]

4. Secondary Outcome: Voucher Utilization Rate
Description: Percent of vouchers utilized by participants in each study arm
Time Frame: Months 1-6 of intervention
Measure: Number (95% Confidence Interval); unit: Percent of vouchers utilized
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
Percent of vouchers utilized | 66.8 [61.6 to 72.0] | 81.8 [76.6 to 86.9] | 67.8 [62.8 to 72.9] | 80.4 [75.4 to 85.5]

5. Other Pre Specified Outcome: Voucher Ease of Use Survey
Description: Survey of how easy participants found it to use vouchers. This is a composite score ranging from 0 (hard) to 3 (easy) based on individual scores of 0 (hard) or 1 (easy) in response to three questions at month 6 (the questions are in the appendix), which assessed participants' understanding of how to use the vouchers, ability to determine which foods were redeemable, and ease of redeeming the voucher with a cashier.
Time Frame: Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
score on a scale | 2.87 [2.75 to 2.99] | 2.72 [2.60 to 2.83] | 2.56 [2.45 to 2.68] | 2.58 [2.47 to 2.69]

6. Other Pre Specified Outcome: Self-reported Height Survey
Description: Self-reported height by phone survey.
Time Frame: Month 6
Measure: Mean (95% Confidence Interval); unit: inches
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
inches | 65.64 [64.70 to 66.57] | 66.03 [65.14 to 66.91] | 66.14 [65.23 to 67.05] | 66.17 [64.43 to 66.91]

7. Other Pre Specified Outcome: Food Security Survey
Description: This is the 6-item United States Department of Agriculture food security scale; the survey questions are in the appendix under "Main Survey." Each of the responses to the 6 questions were scored as a 1 or 0, depending of the particular question. The individual scores were then totaled, and individuals could receive a score anywhere from 0 indicating the most food security to 6 indicating the least food security. Then, the totaled individual 0 to 6 scores (fs_total) were broken into two categories, 0-1 being food secure, and 2-6 being food insecure. The number of participants below reflects the total number of participants who were food secure (that is, scored fs_total = 0-1) at Baseline, Month 6, and Month 12, respectively.
Time Frame: Baseline, Month 6, and Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
Participants
  baseline | 24 | 27 | 37 | 29
  month 6 | 27 | 30 | 42 | 38
  month 12 | 29 | 32 | 31 | 33

8. Other Pre Specified Outcome: Self-reported Weight Survey
Description: Self-reported weight by phone survey.
Time Frame: Month 6
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
Number analyzed (Participants) | 86 | 90 | 92 | 91
pounds | 181.30 [169.67 to 192.93] | 172.77 [163.37 to 182.17] | 178.50 [166.44 to 190.56] | 174.43 [164.63 to 184.23]

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Description: No differences from the clinicaltrials.gov definitions
Arm/Group | 1: Distributed, Targeted Vouchers | 2: Lump Sum, Targeted Vouchers | 3: Distributed, Untargeted Vouchers | 4: Lump Sum, Untargeted Vouchers
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/90 | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/90 | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 0/86 | 0/90 | 0/92 | 0/91

LIMITATIONS AND CAVEATS:
Dietary data are from self-report, via 24-hour dietary recalls. Survey data are from self-reported scales.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02843178/Prot_SAP_ICF_000.pdf